CLINICAL TRIAL: NCT00312988
Title: Topotecan-Monotherapy Vs. Topotecan + Etoposide Vs. Topotecan + Gemcitabine in Therapy in Patients With Recurrent Ovarian Cancer
Brief Title: Topotecan Vs. Topotecan + Etoposide Vs.Topotecan + Gemcitabine in Ovarian Cancer Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031000; Topo Phase III
Record Dates: First submitted 2005-09-09; First posted 2006-04-11 (Estimated); Last update posted 2006-04-11 (Estimated); Status verified 2005-09

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan; Gemcitabine

INTERVENTIONS:
Drug: Hycamtin
Drug: Gemcitabine

SUMMARY:
Determination of total survival under Topotecan Monotherapy, Topotecan + Etoposide and Topotecan + Gemcitabine in second-line therapy in patient with recurrent ovarian cancer.

DETAILED DESCRIPTION:
In Germany ovarian cancer belongs to the most frequently forms of cancer in the female population. The prognosis for women with a platin refractory ovarian cancer is very bad. The median survival time amounts for less a year. Especially in this palliative situation therapies regarding efficacy as well as quality of life are needed. in Germany Topotecan is approved since 1996 for patients after previous treatment with platin, the rare non-hematological side-effects making it interesting for a palliative therapy. Since best results in a chemo-therapeutical treatment are commonly obtained with the combination of two or more cytostatic agents this study tests a Topotecan Monotherapy and two Topotecan combinations. Both combination agents show efficacy alone against solid cancer using from Topotecan different mechanism resulting in different main side effects. Total survival, remission rates, time ti progression and quality of life are the main criteria investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patient with recurrent ovarian cancer
* Second-line chemotherapy
* > = 18 years of age
* ECOG < = 2

Exclusion Criteria:

* ECOG > 2
* Patients with more than one chemotherapy in anamneses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2000-01; Study Completion 2009-12

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
time to progression
determining adverse effects
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Fotopoulou C, Karavas A, Trappe R, Chekerov R, Lichtenegger W, Sehouli J. Venous thromboembolism in recurrent ovarian cancer-patients: A systematic evaluation of the North-Eastern German Society of Gynaecologic Oncology Ovarian Cancer Study Group (NOGGO). Thromb Res. 2009 Nov;124(5):531-5. doi: 10.1016/j.thromres.2009.03.013. Epub 2009 May 8. PMID 19427025
- See also: Related Info — http://www.noggo.de